CLINICAL TRIAL: NCT03926819
Title: A Phase 1 Open Labeled Single Ascending Dose Followed by Multiple Dose Safety and Pharmacokinetic Study of HBI-002 Carbon Monoxide Oral Liquid Drug Product in Healthy Adult Volunteers.
Brief Title: A Study to Assess the Safety and Pharmacokinetics of HBI-002, an Oral Carbon Monoxide Therapeutic, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hillhurst Biopharmaceuticals, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBI-002-001; 2R44HL131065 (NIH)
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Anemia, Sickle Cell
Keywords: Anemia, Sickle Cell; Anemia, Hemolytic, Congenital; Anemia, Hemolytic; Anemia; Hematologic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn; Carbon Monoxide; CO; Heme Oxygenase; HO-1
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Hemolytic, Congenital; Anemia, Hemolytic; Anemia; Hematologic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Ascending Dose (Active Comparator)
  Interventions: Drug: HBI-002
- Multiple Ascending Dose (Active Comparator)
  Interventions: Drug: HBI-002

INTERVENTIONS:
Drug: HBI-002 — Oral liquid carbon monoxide drug product.

SUMMARY:
This is a single center, open label Phase 1 clinical trial in normal adult subjects to assess safety, tolerability, pharmacokinetics, and pharmacodynamics of HBI-002, an orally administered liquid containing carbon monoxide (CO), with single ascending doses (SAD), followed by multiple dose with doses daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Healthy male or female 18-55 years of age inclusive.
3. Negative HBsAg, aHCV, aHIV, and SARS-CoV-2 test.
4. Non-smoker or vaper (no use of tobacco or marijuana products within 3 months of screening).
5. Body weight between 60 kg and 110 kg (inclusive) and with BMI less than 30 kg/m2.
6. Subjects must be healthy as defined by:

   1. absence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic disease, as determined by the Investigator.
   2. liver function: alanine transaminase (ALT) and aspartate transaminase (AST) ≤2 times the upper limit of the normal range
   3. total bilirubin ≤1.5 times the upper limit of the normal range
   4. renal function: creatinine clearance within normal range as assessed by Cockcroft and Gault calculation
   5. carboxyhemoglobin level by venous blood gas ≤ 3.5% (any time prior to the first dose)
   6. venous lactate level <2.0 mmol/L at baseline.
   7. the absence of current clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead ECG, and clinical laboratory tests (hematology and clinical chemistries), as determined by the Investigator.
7. Negative pregnancy tests for females.
8. Subjects must be willing to use a highly effective method of contraception for the duration of the study and for 30 days thereafter.

   1. Male subjects, without a vasectomy, must use a condom and be instructed that their female partner should use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptive, injectable progesterone, subdermal implant or a tubal ligation if the female partner could become pregnant
   2. Female subjects of childbearing potential (not surgically sterilized and less than one year post-menopausal) should use a form of contraception such as an IUD, diaphragm with spermicide, oral contraceptive, injectable progesterone, subdermal implant or a tubal ligation, and be instructed that their male partners should use a condom, if not vasectomized.

Exclusion Criteria:

Subjects who meet any of the following criteria will be ineligible for participation in the study:

1. Subjects with concurrent illness/disease as defined by:

   1. clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic disease, as determined by the Investigator.
   2. current clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead ECG, and clinical laboratory tests (hematology, clinical chemistries and urinalysis), as determined by the Investigator.
   3. clinically significant illness and/or surgery within 4 weeks prior to dosing.
2. Anemia of any cause.
3. Homozygous or heterozygous hemoglobinopathy.
4. Blood transfusion within six weeks prior to the first administration of study drug.
5. Carboxyhemoglobin ≥ 3.5% (any time prior to the first dose)
6. Oxygen saturation by transcutaneous measurement consistently ≤ 95% (any time prior to the first dose)
7. Exposure to any live vaccine within 28 days prior to study drug administration.
8. History of febrile or infective illness within 14 days prior to dosing.
9. Positive pregnancy test or breast feeding for females.
10. Weight loss or gain of more than 5 kg within 3 months prior to dosing.
11. History of alcohol abuse or dependence or regular use of alcohol within six months prior to dosing (defined as more than 14 units of alcohol per week; 1 Unit= 150 mL wine, 360 mL beer or 45 mL of 40% alcohol)
12. Positive result on alcohol screen
13. History of pulmonary infiltrate or pneumonia within 6 months prior to dosing or pulmonary/bronchial infection within 2 weeks prior to dosing.
14. History of cancer, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin more than 1 year prior.
15. History of cardiac disease
16. History of drug abuse or dependence.
17. Positive results on drug screen (oxycodone, benzodiazepines, THC, cocaine, opiates, and methamphetamine).
18. Use of prescription drugs within 7 days or 5 half-lives (whichever is longer) prior to dosing. Herbal and vitamin supplements must be discontinued 14 days prior to dosing.
19. Unwilling or unable to comply with the requirements of the protocol.
20. Treatment with an investigational drug within the longer of 30 days or five half-lives.
21. Systolic blood pressure lower than 90 or above 140 mm Hg, diastolic blood pressure lower than 50 or above 90 mm Hg, heart rate less than 45 or above 100 bpm, or arrhythmia at screening and/or baseline. ECG abnormalities or other vital sign abnormalities that are clinically significant at screening and/or baseline, as determined by the Investigator.
22. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into the study.
23. History of allergic reactions to any of the drug product excipients
24. History of epilepsy or seizure
25. History of suicide attempts or ideation (by medical history)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Company, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Ascending Dose - 0.7 mg/kg; Single Ascending Dose - 1.3 mg/kg; Single Ascending Dose - 2.7 mg/kg; Single Ascending Dose - 3.7 mg/kg: HBI-002: Oral liquid carbon monoxide drug product; adjusted.
- Multiple Dose - 4.4, 3.6, 2.7 mg/kg: HBI-002: Oral liquid carbon monoxide drug product; dosing adjusted to achieve target range.
Period: Overall Study
Arm/Group | Single Ascending Dose - 0.7 mg/kg | Single Ascending Dose - 1.3 mg/kg | Single Ascending Dose - 2.7 mg/kg | Single Ascending Dose - 3.7 mg/kg | Multiple Dose - 4.4, 3.6, 2.7 mg/kg
Started | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SAD - 0.9 mg/kg; SAD - 1.8 mg/kg; SAD - 3.6 mg/kg; SAD - 5.0 mg/kg; Multiple Dose: HBI-002: Oral liquid carbon monoxide drug product.
- Total: Total of all reporting groups
Arm/Group | SAD - 0.9 mg/kg | SAD - 1.8 mg/kg | SAD - 3.6 mg/kg | SAD - 5.0 mg/kg | Multiple Dose | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (8) | 39 (12) | 39 (9) | 38 (7) | 40 (8) | 39 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 2 | 4
  Male | 3 | 4 | 4 | 3 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 1 | 2 | 8
  White | 2 | 0 | 2 | 2 | 2 | 8
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 of dosing, up to 30 days post-dose for SAD cohorts. Day 1 of dosing to 30 days post last dose, up to 37 days for MAD cohort
Measure: Count of Participants; unit: Participants
Groups:
- Single Ascending Dose - 0.9 mg/kg; Single Ascending Dose - 1.8 mg/kg; Single Ascending Dose - 3.6 mg/kg; Single Ascending Dose - 5.0 mg/kg; Multiple Dose: HBI-002: Oral liquid carbon monoxide drug product.
Arm/Group | Single Ascending Dose - 0.9 mg/kg | Single Ascending Dose - 1.8 mg/kg | Single Ascending Dose - 3.6 mg/kg | Single Ascending Dose - 5.0 mg/kg | Multiple Dose
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants
  Serious Adverse Events (SAEs) | 0 | 0 | 0 | 0 | 0
  Severe TEAEs | 0 | 0 | 0 | 0 | 0
  Moderate TEAEs | 0 | 0 | 0 | 0 | 0
  Mild TEAEs | 2 | 1 | 0 | 3 | 3

2. Primary Outcome: Cmax
Description: Maximum COHb Concentration (Cmax), measured by blood gas machine with co-oximetry
Time Frame: Blood samples will be drawn on Day 1 immediately before and after dosing at 30, 60, 90, 120 minutes and at 3, 4, 5, 6, 24, 48, and 72 hours
Measure: Mean (Standard Deviation); unit: percentage COHb saturation
Arm/Group | Single Ascending Dose - 0.9 mg/kg | Single Ascending Dose - 1.8 mg/kg | Single Ascending Dose - 3.6 mg/kg | Single Ascending Dose - 5.0 mg/kg | Multiple Dose
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
percentage COHb saturation | 3.4 (0.1) | 3.8 (0.5) | 5.7 (1.7) | 6.9 (1.6) | 8.7 (1.3)

ADVERSE EVENTS:
Time Frame: Day 1 of dosing, up to 30 days post-dose for SAD cohorts. Day 1 of dosing to 30 days post last dose, up to 37 days for MAD cohort
Arm/Group | SAD - 0.9 mg/kg | SAD - 1.8 mg/kg | SAD - 3.6 mg/kg | SAD - 5.0 mg/kg | Multiple Dose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 0/4 | 3/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD - 0.9 mg/kg (N=4) | SAD - 1.8 mg/kg (N=4) | SAD - 3.6 mg/kg (N=4) | SAD - 5.0 mg/kg (N=4) | Multiple Dose (N=4)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Investigations (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03926819/Prot_SAP_000.pdf